CLINICAL TRIAL: NCT03364270
Title: An Exploratory, Phase II, Open Label, Single-Center, Non-Randomized Study Of [F-18] RGD-K5 Positron Emission Tomography (PET) In Participants With Carotid Artery Stenosis
Brief Title: TRACER [F-18] RDG-K5 Carotid Plaque Imaging Study
Acronym: K5-C200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Balaji Tamarappoo (Other)
Responsible Party: Sponsor-Investigator, Balaji Tamarappoo, Staff, Cardiac Imaging, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00047624
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Carotid Arteries
Keywords: atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — 18F-RGD-K5

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [F-18] RDG-K5 (Experimental): PET/CT Imaging with administration of [F-18] RGD-K5
  Interventions: Drug: PET/CT Imaging with [F-18] RGD-K5

INTERVENTIONS:
Drug: PET/CT Imaging with [F-18] RGD-K5 — PET Imaging/scan with [F-18] RGD-K5, PET Imaging/scan with RGD-K5, PET Imaging/scan with K5
  Other Names: RGD-K5; K5

SUMMARY:
The purpose of this study is to investigate the ability of a new investigational agent compound [F-18] labeled RGD-K5 to detect unstable atherosclerotic plaque in the carotid artery of subjects being considered for carotid endarterectomy (CEA), and to confirm this ability through tissue analysis of samples of carotid artery plaques that will be collected during the planned carotid surgery. [F-18] RGD-K5 is a radioactive tracer used in imaging to detect active growth of new blood vessels and presence of macrophages. Patients with unstable plaque may be prone to rupture of the plaque due to increase in macrophage activity and growth of new blood vessels. [F-18] RGD-K5 is an investigational agent, which means that it has not yet been approved by the US Food and Drug Administration (FDA).

Unstable atherosclerotic plaque that is prone to rupture is characterized by an increase in the number of macrophages and enhanced angiogenesis. Both neovascular endothelium and macrophages exhibit increased Alpha-v beta3 integrin expression. PET (Positron Emission Tomography) imaging of [F-18] RGD-K5 uptake may identify carotid plaque with increased inflammation and neovascularization and may therefore detect unstable plaque in participants with carotid artery stenosis.

Prior to Dr. Tamarappoo's relocation to Cedars Sinai Medical Center (CSMC), 5 subjects were enrolled at the Cleveland Clinic where PET-CT (Positron Emission Tomography - Computed Tomography) was performed. 6 subjects will be scanned at Cedars using PET-MRI (Positron emission tomography-magnetic resonance imaging). Based on preliminary data with PET-CTA, the investigator strongly believes the study will be able to reproducibly detect significant [F-18] RGD-K5 uptake in plaque from symptomatic patients. Ultimately, demonstrating preferential [F-18] RGD-K5 uptake in symptomatic patients will significantly impact the way in which patients with carotid plaque (at risk for stroke) are treated and it may prevent unnecessary surgical and endovascular procedures in this population

DETAILED DESCRIPTION:
The primary objectives of this exploratory study are:

* To assess the uptake of [F-18] RGD-K5 by carotid plaque with PET/MRI imaging in participants prior to carotid endarterectomy and thereby determine if carotid plaque that causes significant stenosis [in participants being considered for carotid endarterectomy (CEA)] is characterized by increased integrin expression and enhanced angiogenesis.
* To collect safety data of [F-18] RGD-K5 in participants with carotid atherosclerosis.

Potential subjects will be identified and approached during an inpatient or outpatient clinical visit by a member of the research team. Potential subjects will be identified by their treating physicians and referred to the researchers. Patients' private and identifiable information will not be shared prior to receiving permission from the patient to do so

Summary of research procedures:

Physical exam and vital Signs:

Height, weight, temperature, heart rate and blood pressure will be checked before beginning the imaging tests. Subjects' heart rate and blood pressure will be checked again after each of the two PET/MRI images, and as needed.

Patients will also be asked about the presence of ICD, pacemaker or any metallic implants that would not be compatible with the MRI magnet (presence of MRI non-compatible devices will be an exclusion criteria)

Blood Test:

If labs have been done and the lab values meet the criteria to participate in this study, the investigators will not need to collect these labs again on the day of testing. If these labs have not been collected within 30 days prior to the research imaging tests, the investigators will draw a tube of blood to check kidney function and other necessary blood values prior to the research testing. Patients with a glomerular filtration rate (GFR) <40ml/min will be excluded from the study.

Urine Pregnancy test:

This will only need to be done in female subjects of childbearing potential. This will need to be checked prior to scheduling subjects' research imaging tests. If subjects' tests are schedules more than 2 days (48 hours) since first checked, this test will need to be rechecked on the day of subjects' research imaging testing.

ECG:

An ECG (electrocardiogram) will be done to assess subjects' heart rhythm before the testing begins, and after each of the PET scans.

IV insertion:

A catheter will be inserted into subjects' arm. It is through this IV catheter that the dose of [F-18] RGD-K5 will be given prior to imaging.

Research PET/MRI Imaging of the Carotid Arteries:

2 hours after receiving the dose of [F-18] RGD-K5 PET/MRI imaging of subjects' neck (carotid arteries) will be performed. Subjects will be lying on subjects' back with a head fixation device supporting subjects' head to prevent Subjects from moving subjects' head while the images are taken. This scan will take about 30-45 minutes. Subjects will be permitted to get up and move around between receiving the radiotracer and imaging. Subjects will be asked to drink a glass of water before receiving the dose of [F-18] RGD-K5.

Histology and Immunohistochemistry:

During Subjects carotid endarterectomy(CEA) which is a clinically indicated procedure, atherosclerotic plaque will be removed. A sample of this plaque will be collected and taken to the histology laboratory at Cedars Sinai for analysis.

Follow Up phone call:

Subjects will be contacted by phone the day after subjects' PET scans to ask if Subjects have had any medical problems and what medications Subjects have taken since the PET scan. If Subjects were seen by a doctor to be evaluated for a medical problem, the investigators may ask permission to contact the doctor or hospital to obtain copies of subjects' medical records

Research poses greater than minimal risk

Anticipated benefits:

There is no personal benefit to participants by participating in this research study.

The knowledge to be gained from this research may be beneficial for other patients, society or science.

The detection by the imaging protocol of unstable atherosclerotic plaque in the carotid artery will not result in any change in their standard of care.

The potential benefit of the study to the patient is that it will allow the physician treating the patient to know the entire extent of the carotid plaque, plaque composition and will inform them of the anatomy of the carotid artery in question.

Furthermore, it will provide information about plaque in the contralateral carotid artery and if that plaque has a high degree of inflammation. If a high inflammatory burden is noted in the contralateral carotid artery, there will be more vigilance in monitoring these patients.

Summary of process by which confidentiality will be maintained:

Research records will be stored in a locked cabinet in a secure location Electronic research records will be stored in a shared network folder on the CSMC network. The list linking the assigned code number to the individual subject will be maintained separately from the other research data. Only certified research personnel who are listed on the approved Institutional Review Board (IRB) application will be given access to identifiable subject information. Research related data and patient/subject information will never be stored on a researcher's personal (private) computer or laptop. Study data will be coded upon abstraction so that Direct Identifiers** are maintained separately from the data set.

Summary of data and safety monitoring plan:

The study will be monitored only by the study investigators and/or sponsor.

How does participation in the research differ from the receipt of standard care:

RISKS OF THE STUDY

As with any research study, there may be adverse events or side effects that are currently unknown and it is possible that certain of these unknown risks could be permanent, serious or life threatening. The study doctor will inform subjects of any significant new information that is discovered during this trial.

Risks of the Study Drug Based upon the toxicity profile to be administered as a single dose, the purity and impurity profile of [F-18] RGD-K5, no risk of adverse events is anticipated for this study.

Radiation Risk:

* It is very unlikely that participants will see any harmful effects because of the radiation exposure participants will receive from taking part in this study.
* At high levels of exposure, scientists agree that radiation can cause cancer. This research study involves exposure to radiation from the RGDK5-PET scan. The total amount of radiation exposure participants will receive is equivalent to a uniform whole-body exposure of 0.8 rem. This is comparable to approximately three years' worth of radiation exposure from typical environmental sources (about 0.3 rem per year, which includes radon, natural background radiation, and cosmic rays). This is also comparable to 16% of the maximum annual exposure for radiation workers (5 rem) allowed by the Nuclear Regulatory Commission.

MRI is not associated with any radiation risk.

MRI non-compatible devices such as pacemakers, ICD (implantable cardioverter defibrillator) and metallic implants may cause artifacts in imaging and device malfunction as well as local tissue injury.

Contrast used for MRI is associated with minimal risk among patients who are free of significant renal dysfunction.

When injected into the body, gadolinium contrast medium makes certain tissues, abnormalities or disease processes more clearly visible on a magnetic resonance imaging scan. They are used to improve the clarity of the scanned images or pictures of the body's internal structures.

Gadolinium contrast medium is given by intravenous injection.

The risk of gadolinium contrast is minimal in patients without severe renal disease.

The most common adverse effects of gadolinium agents are

* Itching of the skin (5%)
* Headache (4%)
* Nausea (4%)
* Very small risk of local pain
* Hypersensitivity (allergic reaction)
* Rarely (<1% of the time) it can cause low blood pressure and lightheadedness. This can be treated immediately with IV fluids.

More serious allergic reactions that are life threatening are rare. Gadolinium is not safe for people with late stage kidney disease or who have had a liver transplant. Gadolinium-based contrast agents increase the risk for a rare, but serious adverse reaction, called nephrogenic systemic fibrosis (NSF) among patients with impaired elimination of the drugs. Patients with kidney disease are at increased risk of developing NSF. NSF may cause skin thickening, joint pain and/or swelling, causing feelings of burning, itching and pain that can be severe. In very rare cases, NSF can lead to lung and heart problems and may be life threatening. Participants will have a blood test to measure kidney function and if the blood test is abnormal, they will not be permitted to receive gadolinium.

There is a very small risk of mild headache and local pain. Rarely (<1% of the time) it can cause low blood pressure and lightheadedness. This can be treated immediately with IV fluids. More serious allergic reactions that are life threatening are rare. Gadolinium is not safe for people with late stage kidney disease or who have had a liver transplant.

As with all research procedures and administration of study drugs, subjects will be monitored at all times.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting

a. to the neurologist for evaluation of stroke or TIA (Symptomatic) with: i. Symptomatic patients with plaque ≥70% in at least one carotid artery that would be implicated as the source of embolus responsible for the stroke/TIA. b. or to the vascular surgeon for CEA (Asymptomatic) with: i. asymptomatic patients with a luminal stenosis of ≥70% in at least one carotid artery (stable plaque) referred for CEA ii. age-matched by deciles to symptomatic patients

Exclusion Criteria:

1. stroke due to atrial fibrillation,
2. preexisting carotid stents in the artery of interest,
3. renal dysfunction defined as glomerular filtration rate (GFR) <40ml/min,
4. allergy to gadolinium based contrast agents,
5. Volunteers who have had four or more prior previous gadolinium contrast scans
6. metal implants incompatible with MRI or other condition that prohibits MRI,
7. pregnancy,
8. inability to provide informed consent and
9. age ≤18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balaji Tamarappoo, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from outpatient clinic or from the hospital.
Groups:
- Patients With Carotid Atherosclerosis: Patients deemed to have carotid artery plaque and with symptoms of stroke or transient ischemic attack or those with significant atherosclerosis defined as >70%.
Period: Overall Study
Arm/Group | Patients With Carotid Atherosclerosis
Started | 6 (First patient to undergo PET-MRI: 10/10/2018)
Completed | 6 (Last subject scanned: 1/9/2020)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Carotid Atherosclerosis: Patients deemed to have carotid artery plaque who had previously experienced symptoms of stroke or transient ischemic attack or those with significant atherosclerosis defined as >70%.
Arm/Group | Patients With Carotid Atherosclerosis
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 66 [62 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Uptake of [F-18] RGD-K5 by Carotid Plaque With PET/MRI Imaging in the Artery Believed to be the Cause of Transient Ischemic Attack (TIA) or Stroke Symptoms Compared to the Contralateral Carotid Artery Not Implicated in TIA or Stroke
Description: To assess the uptake of [F-18] RGD-K5 by carotid plaque with PET/MRI imaging in participants prior to carotid enterectomy and thereby determine if carotid plaque that causes TIA or stroke symptoms is characterized by increased integrin expression and enhanced angiogenesis. Each patient serves as their own control. [F-18] RGD-K5 (radiotracer) uptake is measured (expressed as target to background ratio) in the carotid artery containing the plaque considered responsible for causing stroke or TIA symptoms (culprit plaque).
  Plaque maximum standardized uptake value (RT SUVmax) of the radiotracer is compared to tracer maximum standardized uptake value (RT SUVmax) in the contralateral carotid artery which does not contain cluprit plaque.
Time Frame: within 96 hrs of a stroke or TIA (transient ischemic attack)
Population: We enrolled and imaged with PET-MRI, 6 patients with carotid atherosclerosis. Carotid plaque was imaged 2h post injection of 10-12.5mCi of 18F-RGD peptide. 18F-RGD uptake by atherosclerotic plaque was quantified in the culprit artery implicated in stroke or transient ischemic attack and was compared to 18F-RGD uptake in the contralateral carotid artery.
Measure: Mean (Standard Deviation); unit: Ratio SUV max
Units Other Than Participants: plaque
Groups:
- Arm: Stroke/TIA: Atherosclerotic plaque in the artery implicated in causing stroke or TIA symptoms.
- Arm: Non-Stroke/TIA: 18F-RGD uptake by atherosclerotic plaque in the contralateral artery not implicated in stroke or TIA
Arm/Group | Arm: Stroke/TIA | Arm: Non-Stroke/TIA
Number analyzed (Participants) | 6 | 6
Number analyzed (plaque) | 6 | 6
Ratio SUV max | 1.78 (0.21) | 1.2 (0.15)
Statistical Analysis 1: Comparison: Arm: Stroke/TIA; Null hypothesis: There is no difference in mean 18F-RGD uptake (expressed as a target to background ratio) in the culprit artery (carotid artery implicated in stroke or transient ischemic attack [TIA]) when compared to mean 18F-RGD uptake in the contralateral carotid artery. A paired t-test was used to compare 18F-RGD uptake in culprit plaque to plaque in the contralateral artery; Test type: Other; p = .001, t-test, 2 sided — Threshold p<0.05; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.33 to 0.84]

2. Secondary Outcome: Number of Participants With Carotid Atherosclerosis
Description: To determine if there were any adverse events in patients who underwent PET/MRI imaging with [F-18] RGD-K5.
  We documented and reported the percent of individuals who experienced significant adverse events.
Time Frame: at the time of imaging and immediately following imaging
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Carotid Atherosclerosis: Patients who experienced significant adverse events after undergoing PET-MRI with [18F] RGD-K5 injection.
Arm/Group | Patients With Carotid Atherosclerosis
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: 30 Days
Description: No adverse events were reported.
Arm/Group | [F-18] RDG-K5
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Small sample size Differences in the time between imaging and symptoms of stroke or transient ischemic attack

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03364270/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT03364270/ICF_001.pdf